CLINICAL TRIAL: NCT03665103
Title: Laser-assisted ICSI Effect on Degeneration Rate After ICSI
Brief Title: Laser-assisted ICSI Versus Conventional ICSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Laser-ICSI
Record Dates: First submitted 2018-09-06; First posted 2018-09-11 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser-assisted ICSI (Experimental)
  Interventions: Other: Laser-assisted ICSI
- conventional ICSI (No Intervention)

INTERVENTIONS:
Other: Laser-assisted ICSI — Laser opening of the zona pellucida.
  Arms: Laser-assisted ICSI

SUMMARY:
Degeneration rate after ICSI is expectable but decreasing it is a goal. Laser-assisted ICSI can serve to decrease this degeneration rate.

ELIGIBILITY:
Inclusion Criteria:

* all ICSI cycles

Exclusion Criteria:

* no exclusion

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 966 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
oocyte survival after injection | 6 days of culture

SECONDARY OUTCOMES:
blastocyst formation rate | 6 days of culture
embryo utilization rate | 6 days of culture
clinical pregnancy rate | four weeks after embryo transfer
ongoing pregnancy rate | Twelve weeks of gestation

CONTACTS AND LOCATIONS:
Locations (1):
- IbnSina IVF Center, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fawzy M, Emad M, Mahran A, Abdelrahman MY, Fetih AN, Abdelghafar H, Elsuity MA, Rashed H, Sabry M. A randomized controlled trial of laser-assisted ICSI. Hum Reprod. 2020 Dec 1;35(12):2692-2700. doi: 10.1093/humrep/deaa160. PMID 32995832